CLINICAL TRIAL: NCT02340000
Title: Clinical Trial of the Treatment of Acute Sinusitis With Standard-dose Versus High-dose Amoxicillin/Clavulanate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Paul Sorum, MD, Professor of Internal Medicine and Pediatrics, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3968
Record Dates: First submitted 2014-11-22; First posted 2015-01-16 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Sinusitis
Keywords: acute sinusitis; amoxicillin/clavulanate; adults; outcomes
MeSH Terms: conditions — Sinusitis | interventions — Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard dose (Active Comparator): amoxicillin/clavulanate 875/125 mg + placebo tablet twice a day for 7 days
  Interventions: Drug: standard dose amoxicillin/clavulanate
- high dose (Experimental): Time Period I (November 18, 2014-January 5, 2016): extended-release amoxicillin/clavulanate 1000/62.5 mg 2 tablets (by different manufacturer) twice a day for 7 days Time Period 2 (February 6, 2016-February 27, 2017): immediate-release amoxicillin/clavunate 875/125 mg plus standard immediate-release amoxicillin 875 mg twice a day for 7 days
  Interventions: Drug: high dose amoxicillin/clavulanate

INTERVENTIONS:
Drug: standard dose amoxicillin/clavulanate — amoxicillin/clavulanate 875/125 + placebo bid x 7 days
  Arms: standard dose
Drug: high dose amoxicillin/clavulanate — Time Period I: extended-release amoxicillin/clavulanate 1000/62.5 two tablets bid x 7 days Time Period 2: immediate-release amoxicillin/clavulanate 875/125 plus amoxicllin 875 bid x 7 days
  Arms: high dose

SUMMARY:
The aim is to determine if high-dose amoxicillin/clavulanate is more effective than standard-dose amoxicillin/clavulanate in treating acute bacterial sinusitis in adults seen at a primary care office.

DETAILED DESCRIPTION:
The aim was amended in February 2016--because of the unexpected unavailability of the original high-dose formulation of amoxicillin/clavulanate--to compare the effectiveness (versus standard dose) of extended-release (the original formulation) versus immediate-release amoxicillin/clavulanate.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18 or over
2. Meets definition of acute sinusitis by Infectious Disease Society of America (2012)
3. Clinician and participant chose to start antibiotic treatment

Exclusion Criteria:

1. Previously enrolled in the study
2. Allergic or intolerant to amoxicillin, penicillin, or amoxicillin/clavulanate
3. Specific medication concerns: lactating (since safety of clavulanate unknown); taking allopurinol (increased risk of rash); concurrent mononucleosis (increased risk of rash with amoxicillin); chronic kidney disease with glomerular filtration rate < 30; significant hepatic impairment; history of antibiotic-associated colitis
4. Cognitive impairment so that unable to give informed consent or give reliable assessment of improvement
5. Need to use high-dose amoxicillin/clavulanate: treatment with amoxicllin or penicillin within the past month (risk of penicillin-resistant pneumococci), very ill patient (though not ill enough to send to hospital); immunocompromise
6. Need to hospitalize the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center Internal Medicine and Pediatrics, Latham, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow AW, Benninger MS, Brook I, Brozek JL, Goldstein EJ, Hicks LA, Pankey GA, Seleznick M, Volturo G, Wald ER, File TM Jr; Infectious Diseases Society of America. IDSA clinical practice guideline for acute bacterial rhinosinusitis in children and adults. Clin Infect Dis. 2012 Apr;54(8):e72-e112. doi: 10.1093/cid/cir1043. Epub 2012 Mar 20. PMID 22438350
- [Derived] Matho A, Mulqueen M, Tanino M, Quidort A, Cheung J, Pollard J, Rodriguez J, Swamy S, Tayler B, Garrison G, Ata A, Sorum P. High-dose versus standard-dose amoxicillin/clavulanate for clinically-diagnosed acute bacterial sinusitis: A randomized clinical trial. PLoS One. 2018 May 8;13(5):e0196734. doi: 10.1371/journal.pone.0196734. eCollection 2018. PMID 29738561

RESULTS

PARTICIPANT FLOW:
Period: Time Period 1
Arm/Group | Standard Dose | High Dose
Started | 90 | 89
Completed | 78 | 74
Not Completed | 12 | 15
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Lost to Follow-up | 6 | 7
Period: Time Period 2
Arm/Group | Standard Dose | High Dose
Started | 69 | 67
Completed | 50 | 52
Not Completed | 19 | 15
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Lost to Follow-up | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose | High Dose | Total
Number analyzed (Participants) | 159 | 156 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (15.9) | 45.9 (14.8) | 46.9 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 108 | 223
  Male | 44 | 48 | 92
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Active tobacco use [Count of Participants; unit: Participants] | 19 | 20 | 39
COPD/asthma [Count of Participants; unit: Participants] | 29 | 30 | 59
allergic rhinitis [Count of Participants; unit: Participants] | 82 | 80 | 162
Diabetes [Count of Participants; unit: Participants] | 16 | 15 | 31
Heart disease [Count of Participants; unit: Participants] | 11 | 8 | 19
History of sinusitis [Count of Participants; unit: Participants] | 63 | 60 | 123
Days of illness [Mean (Standard Deviation); unit: days] — Clinician indicated the number of days the patient had been sick prior to the office visit.
  days | 14.8 (8.8) | 14.3 (8.1) | 14.5 (8.4)
Sinusitis category 1 [Count of Participants; unit: Participants] — Duration greater than or equal to 10 days
  Participants | 101 | 103 | 204
Sinusitis category 2 [Count of Participants; unit: Participants] — Severe symptoms (most severe of the 3 categories)
  Participants | 18 | 19 | 37
Sinusitis category 3 [Count of Participants; unit: Participants] — double sickening
  Participants | 40 | 34 | 74
Day 0 SNOT-16 mean item score [Mean (Standard Deviation); unit: units on a scale] — Ratings on a scale from 0=none to 3=severe of 16 sinusitis-related symptoms. Total score can range from 0 to 48 (with 48 the most severe possible)
  units on a scale | 1.89 (.56) | 1.99 (.55) | 1.94 (.55)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Improvement - Day 3 (Rating of "a Lot Better" or "no Symptoms")
Description: rating of "a lot better" or "no symptoms"
Time Frame: end of 3 days of treatment
Population: The number of participants who gave ratings at the end of day 3 of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Standard Dose Time Period I: amoxicillin/clavulanate 875/125 mg + placebo tablet twice a day for 7 days
  standard dose amoxicillin/clavulanate: amoxicillin/clavulanate 875/125 + placebo bid x 7 days
- High Dose Time Period 1: extended-release amoxicillin/clavulanate 1000/62.5 mg 2 tablets twice a day for 7 days
- Standard Dose Time Period 2: Amoxicillin/clavulnate 875/125 plus placebo bid x 7 days
- High Dose Time Period 2: immediate-release amoxicillin/clavunate 872/125 plus amoxicillin 875
Arm/Group | Standard Dose Time Period I | High Dose Time Period 1 | Standard Dose Time Period 2 | High Dose Time Period 2
Number analyzed (Participants) | 87 | 80 | 64 | 63
Participants | 33 | 31 | 22 | 33

2. Secondary Outcome: SNOT-16 - Day 3
Description: Ratings on a scale from 0=none to 3=severe of 16 sinusitis-related symptoms. Total score can range from 0 to 48 (with 48 the most severe possible) of the 16 symptoms.
  The outcome measure was the mean difference in the ratings of each of the 16 symptoms between day 0 and day 3 (values at day 0 minus values at day 3).
Time Frame: day 0, end of 3 days of treatment
Population: The number of participants who gave ratings at day 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard Dose Time Period I: amoxicillin/clavulanate 875/125 mg + placebo tablet twice a day for 7 days
Arm/Group | Standard Dose Time Period I | High Dose Time Period 1 | Standard Dose Time Period 2 | High Dose Time Period 2
Number analyzed (Participants) | 86 | 80 | 62 | 56
units on a scale | .75 (.63) | .87 (.59) | .91 (.63) | .97 (.69)

3. Secondary Outcome: Subjective Improvement - Day 10
Description: rating of "a lot better" or "no symptoms"
Time Frame: end of 10th day
Population: The number of participants who gave a rating at day 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Time Period I | High Dose Time Period 1 | Standard Dose Time Period 2 | High Dose Time Period 2
Number analyzed (Participants) | 78 | 74 | 50 | 52
Participants | 63 | 59 | 35 | 40

4. Secondary Outcome: SNOT-16 - Day 10
Description: Ratings on a scale from 0=none to 3=severe of 16 sinusitis-related symptoms. Total score can range from 0 to 48 (with 48 the most severe possible) of the 16 symptoms.
  The outcome measure was the mean difference in the ratings of each of the 16 symptoms between day 0 and day 10 (values at day 0 minus values at day 10).
Time Frame: day 0, end of 10th day
Population: The number of participants who gave ratings at day 10.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Dose Time Period I | High Dose Time Period 1 | Standard Dose Time Period 2 | High Dose Time Period 2
Number analyzed (Participants) | 79 | 75 | 51 | 53
units on a scale | 1.32 (.71) | 1.48 (.64) | 1.37 (.67) | 1.40 (.73)

5. Secondary Outcome: Nasal Colonization With Resistant Bacteria
Description: Clinicians performed anterior nasal cultures to look for colonization with penicillin-resistant pneumococci and other pathogens (stopped after participant #231 because of lack of funds).
Time Frame: baseline
Population: All 231 participants were analyzed together regardless of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: First 231 participants
Arm/Group | Overall
Number analyzed (Participants) | 231
Participants
  No growth or normal flora | 139
  Methicillin-sensitive Staphylococcus aureus | 32
  Haemophilus influenzae | 25
  Streptococcus pneumoniae | 9
  Moxarella catarrhalis | 9
  Staphylococcus epidermidis | 7
  Methicillin-resistant Staphylococcus aureus | 5

6. Secondary Outcome: Willingness to Take the Study Antibiotic in the Future
Description: whether participants said they would NOT take the antibiotic again
Time Frame: end of 10th day
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Time Period I | High Dose Time Period 1 | Standard Dose Time Period 2 | High Dose Time Period 2
Number analyzed (Participants) | 75 | 74 | 49 | 52
Participants | 8 | 11 | 5 | 8

ADVERSE EVENTS:
Time Frame: 10 days
Description: The number of participants reporting adverse effects was less than the number initially at risk because some patients withdrew before starting treatment or were lost to follow-up for the study. Since they were all patients in our practice, however, we knew--outside of the study---that none of them suffered death or other serious adverse effects.
Arm/Group | Standard Dose Time Period I | High Dose Time Period 1 | Standard Dose Time Period 2 | High Dose Time Period 2
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/89 | 0/69 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/89 | 0/69 | 0/67
Other Adverse Events (participants affected / at risk) | 30/87 | 37/80 | 19/62 | 27/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Time Period I (N=87) | High Dose Time Period 1 (N=80) | Standard Dose Time Period 2 (N=62) | High Dose Time Period 2 (N=57)
Vaginitis (Infections and infestations) | 3 (3) | 11 (11) | 4 (4) | 7 (7) — vaginal itching or discharge at day 3
diarrhea (Gastrointestinal disorders) | 30 (30) | 37 (37) | 19 (19) | 27 (27) — diarrhea at day 3

LIMITATIONS AND CAVEATS:
1. Initial formulation of high-dose amox/clav (extended release) became unavailable, so had to switch after participant #180 to immediate-release.
2. The medical students and residents had trouble reaching some participants for follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-09-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT02340000/Prot_SAP_000.pdf
  • Informed Consent Form (2014-09-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT02340000/ICF_001.pdf